CLINICAL TRIAL: NCT04326842
Title: Optical Coherence Tomography Angiography Evaluation of Ocular Changes in Patients With Carotid Artery Stenosis
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: HZHZS1
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-04

CONDITIONS: Carotid Stenosis
Keywords: Carotid Stenosis; OCTA
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Carotid artery stenosis: Patients with carotid artery stenosis. Procedure: Carotid artery revascularization procedure
  Interventions: Procedure: Carotid artery revascularization procedure; Device: Optical coherence tomography angiography
- Control: Patients without carotid artery stenosis
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Procedure: Carotid artery revascularization procedure — The patients with carotid artery stenosis will be examined before and after finishing the carotid artery revascularization procedure.
  Groups: Carotid artery stenosis
Device: Optical coherence tomography angiography — Examination will be performed using optical coherence tomography angiography. This device allows quantitative analysis, since it provides numerical data about flow area and flow density maps.

SUMMARY:
This study aims to evaluate ocular changes in patients with carotid artery stenosis by optical coherence tomography angiography before and after carotid artery revascularization procedure.

DETAILED DESCRIPTION:
A growing body of research indicates that abnormal ocular microvascular features may serve as a novel biomarker reflecting the severity of underlying cardiovascular, neurodegenerative, and microvascular disease. Since blood flow to the retina is predominantly supplied by the internal carotid artery (ICA), we hypothesized that ocular microvasculature and structure changes may reflect the disease status or therapeutic effects in patients with carotid artery stenosis.

Optical coherence tomography angiography (OCTA) is a novel, non-invasive imaging modality that can be a reliable tool for the qualitative and quantitative assessments of ocular vessels during various ocular pathological or physiological changes. Recent studies have also demonstrated the ability of OCTA to quantify retinal microvascular changes in monitoring cardiovascular risk.

This study aims to evaluate ocular changes in patients with carotid artery stenosis by optical coherence tomography angiography before and after carotid artery revascularization procedure.In this study, the patients with carotid artery stenosis and control group will receive a series of cerebral and ocular examinations including the most important cerebral CT perfusion (CTP) and OCTA. After that, the cerebral and ocular data between the two groups will be compared. Also, the preoperative and postoperative data acquired will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of carotid artery stenosis
* Age-gender-race-matched controls

Exclusion Criteria:

* age <18 years
* intraocular pressure (IOP) >21 mmHg
* VA >logMAR 1.0
* spherical equivalent (SE) between >1.00 or < -6.00 D
* other serious eye diseases which may affect OCTA results including diabetic retinopathy, hypertensive retinopathy, retinal vascular occlusion, age-related macular degeneration, and uveitis
* major intraocular surgery performed in the past 6 months or a history of laser photocoagulation or intravitreal injection
* glaucoma or first-degree relatives with a history of glaucoma; and
* any disease that might cause poor scan quality (image quality <6).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with carotid artery stenosis undergoing cerebral and eye examination and in routine clinical practice will be included
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Huaizhang Shi, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li X, Zhu S, Zhou S, Zhang Y, Ding Y, Zheng B, Wu P, Shi Y, Zhang H, Shi H. Optical Coherence Tomography Angiography as a Noninvasive Assessment of Cerebral Microcirculatory Disorders Caused by Carotid Artery Stenosis. Dis Markers. 2021 Jul 5;2021:2662031. doi: 10.1155/2021/2662031. eCollection 2021. PMID 34326905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carotid Artery Stenosis | Control
Started | 40 | 89
Completed | 31 | 31
Not Completed | 9 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carotid Artery Stenosis | Control | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.68 (6.82) | 55.39 (11.01) | 59.04 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 18 | 27 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Tobacco [Count of Participants; unit: Participants] | 15 | 14 | 29
Alcohol [Count of Participants; unit: Participants] | 11 | 6 | 17
Hypertension [Count of Participants; unit: Participants] | 28 | 21 | 49
Diabetes [Count of Participants; unit: Participants] | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Radical Peripapillary Capillaries Vessel Density
Description: Radical peripapillary capillaries vessel density of Optical Coherence Tomography Angiography（OCTA）
Time Frame: Difference of vessel density in each group at baseline
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis | Control
Number analyzed (Participants) | 31 | 31
percentage of vessel | 55.95 [53.30 to 58.10] | 57.24 [56.00 to 59.20]

2. Primary Outcome: Superficial Vascular Complexes Vessel Density
Description: superficial vascular complexes vessel density of Optical Coherence Tomography Angiography
Time Frame: Difference of vessel density in each group at baseline
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis | Control
Number analyzed (Participants) | 31 | 31
percentage of vessel | 48.65 [45.50 to 51.10] | 52.22 [50.14 to 52.53]

3. Primary Outcome: Deep Vascular Complexes Vessel Density
Description: deep vascular complexes vessel density of Optical Coherence Tomography Angiography
Time Frame: Difference of vessel density in each group at baseline
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis | Control
Number analyzed (Participants) | 31 | 31
percentage of vessel | 49.65 [46.50 to 53.70] | 57.50 [53.80 to 59.85]

4. Primary Outcome: Choriocapillaris Vessel Density
Description: choriocapillaris vessel density of Optical Coherence Tomography Angiography
Time Frame: Difference of vessel density in each group at baseline
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis | Control
Number analyzed (Participants) | 31 | 31
percentage of vessel | 67.41 [62.90 to 69.92] | 68.74 [65.91 to 71.11]

5. Secondary Outcome: Change of Difference of Mean Transit Time(dMTT)
Description: Change of dMTT is the dMTT value at 4 days after carotid artery procedure minus the value at baseline.
  dMTT is that the value of the lesion side minus value of contralateral side. Mean transit time (MTT) corresponds to the average time, in seconds, that red blood cells spend within a determinate volume of capillary circulation.
Time Frame: baseline and 4 days after carotid artery procedure
Population: This Outcome Measure was only assessed in the "Carotid Artery Stenosis" Arm/Group Among the 31 patients in the experimental group, 21 patients had unilateral severe stenosis or occlusion and 7 patients dropped out of the study
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
seconds | -0.22 [-0.46 to -0.16]

6. Secondary Outcome: Change of the Ratio of Cerebral Blood Flow(rCBF)
Description: Change of rCBF is the rCBF value at 4 days after carotid artery procedure minus the value at baseline.
  rCBF is that the CBF value of the lesion side divided by the value of contralateral side.
  CBF refers to the flow of blood through a certain cross-sectional area of cerebrovascular per unit time.
Time Frame: baseline and 4 days after carotid artery procedure
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
ratio | 0.19 [0.02 to 0.31]

7. Secondary Outcome: Changes of Retinal Nerve Fiber Layer
Description: changes of retinal nerve fiber layer of Optical Coherence Tomography Angiography
Time Frame: baseline and 4 days after carotid artery procedure
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
μm | 2.50 [2.00 to 11.00]

8. Secondary Outcome: Changes of Deep Vascular Complexes Vessel Density
Description: changes of deep vascular complexes vessel density of Optical Coherence Tomography Angiography
Time Frame: baseline and 4 days after carotid artery procedure
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
percentage of vessel | 4.00 [0.70 to 6.50]

9. Secondary Outcome: Changes of Radical Peripapillary Capillaries Vessel Density
Description: changes of radical peripapillary capillaries vessel density of Optical Coherence Tomography Angiography
Time Frame: baseline and 4 days after carotid artery procedure
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
percentage of vessel | 1.55 [0.40 to 2.60]

10. Secondary Outcome: Changes of Superficial Vascular Complexes Vessel Density
Description: changes of superficial vascular complexes vessel density of Optical Coherence Tomography Angiography
Time Frame: baseline and 4 days after carotid artery procedure
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage of vessel
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 14
percentage of vessel | 1.70 [0.40 to 2.80]

ADVERSE EVENTS:
Time Frame: 2weeks post-operation
Description: A patient developed cerebral infarction 7 days after operation, which resulted in prolongation of existing hospitalization.
Groups:
- Control: Patients without carotid artery stenosis. Examination will be performed using optical coherence tomography angiography. Control group did not undergo carotid artery surgery.
Arm/Group | Carotid Artery Stenosis | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid Artery Stenosis (N=31) | Control (N=31)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04326842/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT04326842/Prot_SAP_001.pdf